CLINICAL TRIAL: NCT05708690
Title: Topical Application Effect of Tranexamic Acid in Postoperative Bleeding and Blood Products Transfusion After Cardiac Surgery
Brief Title: Topical Effect of Tranexamic Acid in Postoperative Bleeding and Blood Products Transfusion After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dudy Arman Hanafy, Sp. BTKV (K), MARS, Dr.dr.Dudy Arman Hanafy, Sp.BTKV(K)-D, MARS, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRACS; 1706120543 (Other: FKUI - harapan kita national heart center); 1706120530 (Other: FKUI - harapan kita national heart center)
Record Dates: First submitted 2023-01-09; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease; Surgical Blood Loss
Keywords: CABG; OPCAB; Heart Valve Surgery; Tranexamic Acid; Postoperative Bleeding; Blood Product Transfusion
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: A double-blind, single center, parallel phase 4 randomized clinical trial was conducted with two intervention arms: an intervention arm with the use of tranexamic acid topical and a control arm with the use of normal saline in which the subjects' recruitment and treatment were conducted simultaneously by means of a block randomization.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects were not aware of the arms/treatment given as they were under general anesthesia during the application of interventions being studied. Besides, during the informed consent for the elective cardiac surgery, subjects were extensively given explanation of the purpose, methods, benefits and risks of the procedure including the randomized nature of the allocation to either arms of the study.
  Principal investigators as well as outcomes assessor were kept unaware of the randomization of interventions as they both were restricted for assessing the patients' medical record and the patient identity were coded in the primary database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid Topical (Experimental): The treatment of interest was application of Topical Tranexamic Acid (5 gram in 50 mL warm normal saline). The topical will be poured into the pericardial and mediastinal cavities (after protamine administration), and sternum (before chest closure)
  Interventions: Drug: Tranexamic Acid 100 MG/ML
- Placebo (Placebo Comparator): The control group is given 100 mL of warm normal saline. The topical will be poured into the pericardial and mediastinal cavities (after protamine administration), and sternum (before chest closure).
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — Tranexamic acid is a synthetic derivative of lysine used as an antifibrinolytic in the treatment and prevention of major bleeding. Tranexamic acid competitively and reversibly inhibits the activation of plasminogen via binding at several distinct sites, including four or five low-affinity sites and one high-affinity site, the latter of which is involved in its binding to fibrin. The binding of plasminogen to fibrin induces fibrinolysis - by occupying the necessary binding sites tranexamic acid prevents this dissolution of fibrin, thereby stabilizing the clot and preventing hemorrhage
  Other Names: Tranexamic Acid
  Arms: Tranexamic Acid Topical
Drug: normal saline — Normal saline is a cornerstone of intravenous solutions commonly used in the clinical setting. It is a crystalloid fluid administered via an intravenous solution. Its indications include both adult and pediatric populations as sources of hydration and electrolyte disturbances
  Arms: Placebo

SUMMARY:
This is a single-center, double-blind, randomized controlled trial (RCT) comparing two groups of application of topical dose of tranexamic acid (TxA) versus placebo in patients undergoing coronary artery bypass graft (CABG), off pump coronary bypass graft cardiac surgery (OPCAB), and adult heart valve surgery. The primary outcomes of this study comprised of two parameters; post operative bleeding and blood product transfusion. The primary outcomes were assessed during the operation, until 48-hour post operative.

DETAILED DESCRIPTION:
A single center randomized controlled trial (RCT) was conducted at Harapan Kita National Cardiovascular Center, Jakarta, Indonesia as the tertiary cardiovascular referral hospital. The RCT was conducted from October 1 th, 2022 until January 6 th, 2023 (current status: completed). This study aims to determine whether topical tranexamic acid is more effective on the amount of bleeding and the need for postoperative blood product transfusion compared with placebo in patients undergoing cardiac surgery and specifically measure the difference outcome between coronary artery bypass graft (CABG), off pump coronary bypass graft cardiac surgery (OPCAB), and adult heart valve surgery. The control group in this study is given 100 mL of normal saline. The subjects were adults undergoing elective cardiac surgery (CABG, OPCAB, and heart valve surgery). Both the patients and the principal investigators were blinded for the treatment-control allocation. The patients were purposively selected and were randomly assigned to one of the arms with block randomization. The primary outcomes of this study comprised of two parameters; post operative bleeding and blood product transfusion. The primary outcomes were assessed during the operation, until 48-hour post operative.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages > 18 years old
* Patients who are scheduled electively for cardiac surgery in National Heart Center Harapan Kita, Jakarta, Indonesia
* Patients with heart valve disease indicated for aortic or mitral repair/replace
* Patients with coronary artery disease indicated for CABG or OPCAB surgery
* Aortic and/ mitral valve surgery concomitant with tricuspid repair
* Patients who are agreed to participate in this study

Exclusion Criteria:

* Not willing to become research subjects
* Allergy to tranexamic acid
* Undergoing minimally invasive surgery
* Undergoing double valve (aorta & mitral) procedure and double procedure (CABG+valve, valve+maze)
* Emergency surgery
* History of bleeding disorder or coagulopathy
* History of thromboembolic or hemorrhagic disease
* Active Infective endocarditis
* History of previous cardiac surgery
* Estimated glomerular filtration rate <30 mL/min or on dialysis
* Receiving oral therapy with clopidogrel, aspirin, dabigatran, or rivaroxaban in the last five days
* Receiving chronic warfarin therapy who have not stopped their medication and have an international normalized ratio (INR) >1.5 before surgery
* Pre-operative thrombocytopenia (<50,000 platelets per µL)
* Pregnancy or breast feeding
* Refusal of blood products
* Pericarditis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Initial Postoperative bleeding | immediately after the surgery
  The study parameter is assessed by postoperative chest tube production immediately after the surgery
6-hour postoperative bleeding | within 6-hour after the surgery
  The study parameter is asses the accumulation of drain production within 6 hours postoperatively after surgical procedure
24-hour postoperative bleeding | within 24-hour after the surgery
  The study parameter is asses the accumulation of drain production within 24 hours postoperatively after surgical procedure
48-hour postoperative bleeding | within 48-hour after the surgery
  The study parameter is asses the accumulation of drain production within 48 hours postoperatively after surgical procedure
Postoperative blood product transfusion | participants will be followed for the duration of ICU and intermediate ward stay, an expected average of 5-7 days
  The amount of red blood cell, fresh frozen plasma, thrombocyte concentrate, and cryoprecipitate transfusions the patient receive postoperatively during their stay in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Komite Etik Pusat Jantung Nasional Harapan Kita, Study Chair — Ethical Committee of National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
the study protocol, ethical clearance letter, the primary database of the study, as well as the study's analysis plan and the manuscript of the study will be made available on the permission by the grant provider and ethical committee
Supporting Information: Study Protocol, ICF, CSR
Time Frame: January 6, 2022 for 2 (two) years
Access Criteria: for peer-reviewing or for further analysis or when needed by authors of a systematic review/meta analysis of randomized controlled trials

REFERENCES:
- [Background] Ausen K, Pleym H, Liu J, Hegstad S, Nordgard HB, Pavlovic I, Spigset O. Serum Concentrations and Pharmacokinetics of Tranexamic Acid after Two Means of Topical Administration in Massive Weight Loss Skin-Reducing Surgery. Plast Reconstr Surg. 2019 Jun;143(6):1169e-1178e. doi: 10.1097/PRS.0000000000005620. PMID 31136475
- [Background] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Result] Habbab LM, Hussain S, Power P, Bashir S, Gao P, Semelhago L, VanHelder T, Parry D, Chu V, Lamy A. Decreasing Postoperative Blood Loss by Topical vs. Intravenous Tranexamic Acid in Open Cardiac Surgery (DEPOSITION) study: Results of a pilot study. J Card Surg. 2019 May;34(5):305-311. doi: 10.1111/jocs.14027. Epub 2019 Mar 25. PMID 30908754
- [Result] Abul-Azm A, Abdullah KM. Effect of topical tranexamic acid in open heart surgery. Eur J Anaesthesiol. 2006 May;23(5):380-4. doi: 10.1017/S0265021505001894. Epub 2006 Jan 27. PMID 16438759
- [Result] Baric D, Biocina B, Unic D, Sutlic Z, Rudez I, Vrca VB, Brkic K, Ivkovic M. Topical use of antifibrinolytic agents reduces postoperative bleeding: a double-blind, prospective, randomized study. Eur J Cardiothorac Surg. 2007 Mar;31(3):366-71; discussion 371. doi: 10.1016/j.ejcts.2006.12.003. Epub 2007 Jan 10. PMID 17218108

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT05708690/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT05708690/ICF_001.pdf